CLINICAL TRIAL: NCT03494972
Title: A Tetracycline Drain Reduces Alveolar Osteitis in Third Molar Surgery
Acronym: Wisdomsteeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Tore Bjornland, Professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2015/2168/REK sør-øst B
Record Dates: First submitted 2018-04-04; First posted 2018-04-11 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Post-Operative Wound Infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- drain (Active Comparator): Tetracyclin drain
  Interventions: Drug: Tetracyclin ointment
- No-drain (Sham Comparator): No drain
  Interventions: Drug: Tetracyclin ointment

INTERVENTIONS:
Drug: Tetracyclin ointment — During 3rd molar surgery

SUMMARY:
The aim of this study was to investigate the effect of an oxytetracycline impregnated gauze drain on the incidence of alveolar osteitis (AO) and postoperative pain during the first week after mandibular third molar surgery.

DETAILED DESCRIPTION:
The study was designed as a single-blinded randomized controlled trial. Patients were randomized in two groups by a sealed envelope system: a drain group and a control group. The study population comprised patients undergoing surgical removal of one or both mandibular third molars (3M) during January 2016 until March 2017. Patients referred to our department, who fulfilled the inclusion criteria, were asked to participate in the study. Patients were prospectively included after giving written informed consent.

The inclusion criteria were: age >18 years, indication for removal of one or both 3M, ASA I-II, no need for sedatives, possession of a smartphone with internet access (to be able to register pain score and use of analgesics, see "Data collection methods and statistical analysis"), and being able to attend a postoperative examination after 1 week. Exclusion criteria were: age <18 years, no indication for removal of 3M, ASA III or higher, pregnancy or breastfeeding, need for sedatives or systemic antibiotics, not possessing a smartphone, and not being able to attend a postoperative examination after 1 week. The National Institutes of Health's Consensus Statement (1979) and the American Association of Oral and Maxillofacial Surgeons White Paper on Third Molar Data (2007) served as guidelines when evaluating indication for 3M removal (NIH Consensus Statement 1979, AAOMS White Paper 2007).

Study population (n=200) and group size (n=100) were determined through power analysis: 90% power, 5% significance level and an expected difference of up to 10% between the two groups.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria were: age >18 years, indication for removal of one or both 3M, ASA I-II, no need for sedatives, possession of a smartphone with internet access (to be able to register pain score and use of analgesics, see "Data collection methods and statistical analysis"), and being able to attend a postoperative examination after 1 week.

Exclusion Criteria:

Exclusion criteria were: age <18 years, no indication for removal of 3M, ASA III or higher, pregnancy or breastfeeding, need for sedatives or systemic antibiotics, not possessing a smartphone, and not being able to attend a postoperative examination after 1 week.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-01-02 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Alveolar ostitis | One week
  Registration of pain

CONTACTS AND LOCATIONS:
Overall Officials: Tore Bjornland, PhD, Principal Investigator — Chair Dep oral Surgery and Oral Medicine
Locations (1):
- Tore Bjornland, Oslo, Norway